CLINICAL TRIAL: NCT07314996
Title: A Randomized Controlled Trial of Laparoscopic Versus Open Surgery for Colon Cancer With Visceral Obesity
Brief Title: Laparoscopic Versus Open Surgery for Colon Cancer With Visceral Obesity
Acronym: LOVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jun Li, Chief, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZhejiangU Jun Li
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Colonic Neoplasms
Keywords: laparoscopic surgery; open surgery; Body Round Index (BRI); complete mesocolic excision; oncologic outcome; specimen quality
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy; Conversion to Open Surgery

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned in a 1:1 ratio to undergo laparoscopic surgery or open surgery. Both groups adhered to the principles of Complete Mesocolic Excision (CME), with at least D2 lymph node dissection performed. For patients with suspected mesenteric lymph node metastasis detected by preoperative CT, D3 lymph node dissection was feasible. The intestinal segments 10 cm or more proximal and distal to the tumor were resected.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Surgery Group (Active Comparator): The abdominal cavity is insufflated to establish a pneumoperitoneum for surgical exposure, and laparoscopic surgery is initiated by inserting the laparoscope through a trocar site into the peritoneal cavity.
  Laparoscopic intracorporeal anastomosis is feasible. The specimen must be retrieved through an abdominal wall incision. The dissection sequence is determined by the surgeon's preference.
  Interventions: Procedure: Laparoscopic surgery
- Open Surgery Group (Experimental): Open surgery involves making an abdominal incision to dissect through the skin, subcutaneous tissue, fascia, and muscle, thereby accessing the peritoneal cavity and enabling direct manual manipulation of intra-abdominal organs for surgical intervention.
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — It refers to the scenario where the necessary anatomy for colon cancer resection is performed using laparoscopic instruments. In laparoscopic surgery, conversion to open surgery is defined as making an abdominal wall incision before completing the predetermined necessary anatomical dissection.This study does not permit the use of hand-assisted laparoscopic surgery, single-port laparoscopic surgery, or robotic surgery. The surgery will be performed according to standards of Complete Mesocolic Excision (CME).
  Arms: Laparoscopic Surgery Group
Procedure: Open surgery — It refers to a surgical procedure where the surgeon enters the abdominal cavity through an abdominal wall incision, gains adequate surgical space, and performs anatomical dissection under direct visual guidance, without relying on pneumoperitoneum or laparoscopic camera assistance.
  Arms: Open Surgery Group

SUMMARY:
This study aims to elucidate whether there is a difference in long-term prognosis between laparoscopic surgery and open surgery in colon cancer patients with visceral obesity.

DETAILED DESCRIPTION:
Study on Surgical Approaches for Colon Cancer Patients with Visceral Obesity

Colorectal cancer stands as a major malignant tumor threatening human health. Laparoscopic surgery has been widely adopted in colon cancer treatment, as it yields comparable survival outcomes to open surgery while offering the advantage of minimal invasiveness. However, with the global escalation of obesity, laparoscopic intervention becomes increasingly challenging in colon cancer patients with visceral obesity, potentially compromising surgical quality.

Notably, earlier landmark studies including COST, COLOR, and CLASICC have confirmed that laparoscopic surgery is non-inferior to open surgery in colon cancer patients. Nevertheless, these studies enrolled relatively lean patients with a Body Mass Index (BMI) below the average level of their respective regions; the COLOR study even excluded patients with a BMI exceeding 30 kg/m². Additionally, transverse colon cancer and splenic flexure colon cancer were excluded from these trials, rendering their data insufficiently representative of the growing population of obese colon cancer patients.

In contrast, the JCOG0404 study specifically demonstrated that colon cancer patients with a BMI ≥ 25 kg/m² had significantly poorer prognostic outcomes after laparoscopic surgery compared to open surgery. Further evidence from European waist-to-hip ratio studies and meta-analyses indicates that obese patients-especially those with abdominal obesity-pose greater surgical challenges. For such patients, laparoscopic surgery is associated with fewer harvested lymph nodes, higher conversion rates to open surgery, and potentially compromised surgical quality, which may ultimately lead to inferior long-term prognosis.

The Body Round Index (BRI), calculated using height and waist circumference, serves as a robust predictor of Visceral Fat Area (VFA). It exhibits superior performance to traditional anthropometric indicators such as BMI, waist circumference, and waist-to-hip ratio. Based on BRI and BMI data from Chinese and American populations, as well as clinical observations by the research team, patients with a BRI ≥ 5.0 present with significant visceral fat accumulation, which substantially increases the complexity of surgical procedures.

This study is designed as a prospective, international, multicenter, randomized, open-label, parallel-controlled trial to clarify whether open surgery is superior to laparoscopic surgery in terms of long-term outcomes for colon cancer patients with visceral obesity (defined as BRI ≥ 5.0). Eligible participants meeting all inclusion criteria will be enrolled and randomly assigned in a 1:1 ratio to either the laparoscopic surgery group or the open surgery group. Both groups will undergo surgery adhering to the Complete Mesocolic Excision (CME) standard. Postoperatively, patients will be followed up for 5 years in accordance with the predefined follow-up protocol. The primary outcome measure is the 3-year disease-free survival rate, while secondary outcomes include specimen quality, 30-day postoperative complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Body Roundness Index (BRI) ≥ 5.0, with no laparoscopic surgery contraindications as assessed by the surgeon;
2. Pathologically confirmed colon adenocarcinoma, mucinous adenocarcinoma, or signet ring cell carcinoma;
3. Tumor lower edge > 12 cm from the anus as measured by colonoscopy, and the tumor lower edge not directly palpable by digital rectal examination;
4. Single primary lesion;
5. Aged 18 (inclusive) to 75 (inclusive) years;
6. Clinical stage T3/4Nany or T1-4N+ on chest non-contrast CT and abdominal enhanced CT, no distant metastasis, and resectable as judged by the surgeon;
7. Treatment-naive, no prior anti-tumor treatment;
8. Completed blood routine, liver and kidney function tests, carcinoembryonic antigen (CEA), and carbohydrate antigen 199 (CA199) before randomization, with American Society of Anesthesiologists (ASA) score ≤ III;
9. Patient able to understand the study protocol and willing to participate in the study.

Exclusion Criteria:

1. Height and waist circumference data are unavailable;
2. Hereditary colorectal cancer (Lynch syndrome or Familial Adenomatous Polyposis [FAP]);
3. History of previous malignant neoplasm, with the exception of basal cell carcinoma/papillary thyroid carcinoma/various types of in situ cancers/micro-invasive early-stage lung cancer;
4. Acute exacerbation of major organ diseases (such as, but not limited to, COPD, coronary heart disease, and renal insufficiency) and/or severe acute infectious diseases (such as, but not limited to, hepatitis, pneumonia, and myocarditis);
5. The tumor presents with obstruction or is at high risk of obstruction, and/or there is bleeding and/or perforation, which may necessitate emergency surgery;
6. Pregnancy or breastfeeding;
7. Inability to undergo contrast-enhanced CT scan;
8. Additional surgery after EMR or ESD;
9. Patients with unremitted severe mental illness, moderate or above cognitive impairment (MMSE ≤ 23 points), or those who have been hospitalized due to mood disorders in the past year or have unstable antipsychotic medication;
10. Patients with enlarged mesenteric root lymph nodes detected by preoperative CT or intraoperative exploration and suspected metastasis, or suspected metastasis in organs such as peritoneum or liver detected by intraoperative exploration;
11. Patients with a history of major abdominal surgery and severe adhesions precluding laparoscopic surgery upon laparoscopic exploration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Three-year disease-free survival (DFS) | 36 months post-randomization
  Disease free survival（DFS）was defined as the time from randomization to the first occurrence of locoregional recurrence, distant metastasis, any new primary cancer, or death from any cause

SECONDARY OUTCOMES:
Length of colon resected | 2 weeks post operation.
  Follow the criteria described by Professor Quirke's criteria (BJS 2014, PMID: 25139143)
Length of small bowel resected | 2 weeks post operation.
  Limited to right hemicolectomy. Follow the criteria described by Professor Quirke's criteria (BJS 2014, PMID: 25139143)
Distance between tumor and closest arterial vascular division | 2 weeks post operation.
  Follow the criteria described by Professor Quirke's criteria (BJS 2014, PMID: 25139143)
Distance between nearest bowel wall and the same vascular division | 2 weeks post operation.
  Follow the criteria described by Professor Quirke's criteria (BJS 2014, PMID: 25139143)
Area of mesentery resected | 2 weeks post operation.
  Follow the criteria described by Professor Quirke's criteria (BJS 2014, PMID: 25139143)
Mesocolic grading | 2 weeks post operation.
  Follow the criteria described by Professor West's criteria (Lancet Oncol 2008，PMID: 18667357). This classification system includes three grades: Mesocolic plane, Intramesocolic plane, Muscularis propria plane.
Number of lymph nodes harvested | 2 weeks post operation.
  Follow the criteria described by Professor Quirke's criteria (BJS 2014, PMID: 25139143)
Incidence of intraoperative complications | From the start of surgical skin incision to the completion of skin suturing.
  Intraoperative complications refer to accidents that occur during surgery. Complications may cause harm to the patient or threaten their life safety (such as iatrogenic intestinal injury, vascular injury or other organ injuries, severe bleeding, cardiovascular and cerebrovascular events or respiratory dysfunction that lead to the interruption of surgery, etc.). These events may result in the prolongation of the surgery, changes in the surgical method, unplanned medical interventions, or even endanger the patient's life.
  The study provides classifications and definitions of common complications. For complications not included in the classification table, refer to the Common Terminology Criteria for Adverse Events (CTCAE) V6.0.
Incidence 30-day postoperative complications | From the completion of skin suturing to 30 days after surgery.
  Postoperative complications refer to symptoms and signs diagnosed through imaging or clinical evaluation after surgery .
  The study provides classifications and definitions of common complications. For complications not included in the classification table, refer to the Common Terminology Criteria for Adverse Events (CTCAE) V6.0.

OTHER OUTCOMES:
Quality of life of patients | The survey time points included: preoperatively, 5 days postoperatively, 1 month postoperatively, and 12 months postoperatively.
  The EORTC QLQ-C30 scale was adopted. The corresponding language version was selected according to the patient's place of origin.
Incidence of postoperative abdominal wall incisional hernia | 24-36 months postoperatively
  Diagnostic criteria: The surgical incision area in this study is characterized by an abdominal wall defect with abdominal contents protruding outward through the defect; physical examination shows a significant bulging of the hernia mass when standing or when abdominal pressure increases (e.g., coughing, breath-holding), and the hernia mass can spontaneously reduce when lying down (excluding incarcerated/strangulated incisional hernias). The above lesions must be clearly confirmed by abdominal computed tomography (CT) examination (including three-dimensional reconstruction). （Guidelines for diagnosis and treatment of abdominal wall incision hernia (2024 edition), PMID: 39794142）
5-year overall survival rate | 5 years from randomization.
  The proportion of patients who survived 5 years from randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the requirements of the International Committee of Medical Journal Editors, the de-identified raw data of this study will be made public after the results are published. The access method will be stated when the research results are published.
Supporting Information: Study Protocol, SAP
Time Frame: The access method will be stated when the research results are published.
Access Criteria: To access the Individual Participant Data (IPD), a detailed data usage plan must be submitted, specifying the research objectives and study content, which will be approved following review by the Principal Investigator (PI) of this study.
URL: https://icstac.com.cn/coopCourse?pid=2

REFERENCES:
- See also: WHO acceleration plan to stop obesity. Updated July 3, 2023. — https://www.who.int/publications/i/item/9789240075634
- See also: Mean body mass index trends among adults, age-standardized (kg/m²) Estimates by country by WHO. — https://apps.who.int/gho/data/view.main.CTRY12461?lang=en